CLINICAL TRIAL: NCT04079959
Title: Endometrial Leucocytes Around the Time of Embryo Implantation in Women Undergoing in Vitro Fertilization- Embryo Transfer (IVF-ET)
Brief Title: Endometrial Leucocytes Around the Time of Embryo Implantation in Women Undergoing in IVF-ET
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Chen Xiaoyan, Research Assistant Professor, Chinese University of Hong Kong
Other Study IDs: 2019.277
Record Dates: First submitted 2019-08-27; First posted 2019-09-06 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Pregnancy Related

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — endometrial samples will be stored
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- women who are undergoing frozen embryo transfer: endometrial biopsy will be done one cycle before the frozen embryo transfer
  Interventions: Procedure: endometrial biopsy

INTERVENTIONS:
Procedure: endometrial biopsy — . Endometrial samples are obtained using a biopsy catheter as follows: the Pipette is inserted through the cervical os and advanced gently until resistance is felt. The inner piton of the device is then withdrawn to create suction, and the endometrial sample is obtained by moving the pipette up and down approximately 2-3 cm within the uterine cavity. The device is rotated 360° to ensure adequate coverage of the area.

SUMMARY:
Uterine natural killer (uNK) cells have been implicated to play a role in female reproductive performance. Serval studies showed an increased uNK cell density in the endometrium of women with reproductive failure. In this study, we wish to investigate the density and clustering of four different immune cells.

DETAILED DESCRIPTION:
Implantation is a process whereby the embryo attaches itself to the endometrium. In humans, the endometrium has a specific period of uterine receptivity, which occurs 5-7 days after ovulation and remains receptive for ~4 days (cycle days 20-24), when embryo implantation starts. Implantation failure refers to the failure of the embryo to reach a stage when intrauterine gestational sac is recognized by ultrasonography. It occurs when the embryo is abnormal or when endometrial function is impaired.

Uterine natural killer (uNK) cells have been implicated to play a role in female reproductive performance. They comprise 70-80% of the total leukocyte population in the endometrium during implantation and early pregnancy. Several studies showed an increased uNK cell density in the endometrium of women with reproductive failure. To better understand the contribution of various immune factors to endometrial function and future pregnancy, it is proposed to examine the major immune cells in the same specimen to measure the relative magnitude of the cell density changes and the degree of clustering between two immune cell types.

The aim of this study is to investigate the endometrial leucocytes profile around the time of embryo implantation.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing frozen embryo transfer.

Exclusion Criteria:

* Women older than 40 years
* Women who have any uterine anomaly or intrauterine pathology such as:

Endometrial polyp or/ and Large fibroid with a diameter >4 cm

* Visible hydrosalpinx on transvaginal ultrasound scans
* BMI >35

Ages: 18 Years to 40 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — Endometrial biopsies will be collected for all the participants
Study Population: Women undergoing frozen embryo transfer.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2019-09-15 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
immune cell counting | up to 2 months
  The counting method will be performed according to an agreed and published standardized protocol by a multicenter working group designed to reduce variance of results between centres. Ten images of 40X magnification fields will be analyzed for each sample. The first field to be captured should be selected at random, ensuring that it contained the luminal epithelial border. Subsequent fields should be obtained by moving one field to the left or right of the original field, keeping the luminal epithelial border in view.
Quantification of endometrial immune cells spatial distribution | up to 2 months
  In each 200 times under the microscope vision, based on the X and Y position of each single cell which InForm system could provide, the relative spatial distribution of each individual endometrial immune cell will be considered as a bivariate point pattern

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoyan Chen, PhD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided
Please contact the principle investigator if there is any enquiry